CLINICAL TRIAL: NCT02635347
Title: Remote Ischemic Conditioning (RIC) in Recipients of Brain Death Donor Livers - A Feasibility and Safety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Baburao Koneru, MD, MPH, Professor, Department of Surgery, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro20150002276
Record Dates: First submitted 2015-12-06; First posted 2015-12-18 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-07

CONDITIONS: Liver Failure; Carcinoma, Hepatocellular
Keywords: Remote ischemic preconditioning; Remote ischemic perconditioning; Remote ischemic postconditioning; Remote ischemic conditioning; Orthotopic liver transplant; Brain Death Organ Donor
MeSH Terms: conditions — Liver Failure; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remote Ischemic Conditioning (RIC) group (Experimental): Participants will receive RIC during transplant and the initial four post-transplant days. During transplant: first intervention after induction of anesthesia but before commencing surgery and the second at the conclusion of the procedure. After transplant: RIC applied daily during the first four consecutive postoperative days. Pneumatic tourniquet will be used to induce RIC
  Interventions: Procedure: Remote Ischemic Conditioning (RIC); Device: Pneumatic tourniquet

INTERVENTIONS:
Procedure: Remote Ischemic Conditioning (RIC) — Each RIC intervention will comprise three cycles of 5 minutes of inflation followed by 5 minutes of deflation of a pneumatic tourniquet placed in mid-thigh.
Device: Pneumatic tourniquet — Portable Tourniquet System(PTSii, Delfi Medical Innovations, Inc.) used to perform RIC interventions.

SUMMARY:
This study will assess the feasibility of lower limb-ischemia induced Remote Ischemic Conditioning (RIC) in the perioperative period before, during, and after Orthotopic Liver Transplantation (OLT). Remote ischemic conditioning will consist of 3 cycles of 5 minutes of lower limb ischemia induced via a mid-thigh pneumatic tourniquet, followed by 5 minutes of reperfusion. Interventions will take place after anesthesia induction but before surgery, at the completion of the procedure, and on the mornings of post-operative days 1-4.

DETAILED DESCRIPTION:
Orthotopic liver transplantation (OLT) is associated with a very high risk of complications. In a recent multi-center study of 450 patients, 79% had at least one complication and 63% had severe (Clavien-Dindo grade III or higher) complications. The number and severity of complications are associated with death within 30 days, hospital length of stay, graft and patient survival. Infections are the most common group of complications, followed by pulmonary, renal and liver graft dysfunction. Interventions that decrease these complications after OLT are likely to improve clinical outcomes.

Remote ischemic conditioning is an innate biological phenomenon wherein a brief single or repetitive ischemic stimulus in an organ or tissue such as skeletal muscle induce protection in remote/distant organs against ischemia and other noxious stimuli. This effect can be induced by inflating a pneumatic tourniquet on a leg or arm for a few minutes (usually 5-10) and subsequently deflating to allow reperfusion. This process is usually repeated 3-4 times to ensure an adequate dose of the conditioning stimulus. The conditioning stimulus could be applied before (Preconditioning), concurrent with (Perconditioning), or soon after the index noxious/ischemic insult (Postconditioning).

The goal of this study is to assess the feasibility, patient acceptance, and safety of RIC in liver recipients. In addition, the investigators will obtain data on posttransplant complications. Information obtained from this study will help guide the design of a future randomized, controlled trial to test the benefit of RIC in liver recipients.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years of age) with acute and chronic liver failure requiring liver transplants or patients undergoing transplantation for hepatocellular carcinoma.
* Both sexes
* Written consent to participate in the study

Exclusion Criteria:

* < 18 years of age
* Recipients of split livers
* Retransplantation
* Recipients of livers combined with other organs
* Recipients of livers from cardiac death donors
* Lower extremity amputees
* History of peripheral vascular disease
* Patients taking sulfonylurea anti-diabetic agents at the time of transplant
* Patients taking nitrates at the time of transplant
* Body mass index > 45
* Pregnant patients
* Patients in whom complete lower extremity ischemia is not achieved despite maximum tourniquet inflation to 250 mmHg during the first intervention
* Patients with lower extremity paralysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-11; Primary Completion 2017-10-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baburao Koneru, MD, MPH, Principal Investigator — Rutgers University
Locations (1):
- Rutgers University - University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parikh A, Washburn KW, Matsuoka L, Pandit U, Kim JE, Almeda J, Mora-Esteves C, Halff G, Genyk Y, Holland B, Wilson DJ, Sher L, Koneru B. A multicenter study of 30 days complications after deceased donor liver transplantation in the model for end-stage liver disease score era. Liver Transpl. 2015 Sep;21(9):1160-8. doi: 10.1002/lt.24181. PMID 25991395
- [Background] Huang CT, Lin HC, Chang SC, Lee WC. Pre-operative risk factors predict post-operative respiratory failure after liver transplantation. PLoS One. 2011;6(8):e22689. doi: 10.1371/journal.pone.0022689. Epub 2011 Aug 1. PMID 21829646
- [Background] Levesque E, Hoti E, Azoulay D, Honore I, Guignard B, Vibert E, Ichai P, Antoun F, Saliba F, Samuel D. Pulmonary complications after elective liver transplantation-incidence, risk factors, and outcome. Transplantation. 2012 Sep 15;94(5):532-8. doi: 10.1097/TP.0b013e31825c1d41. PMID 22885879
- [Background] Gracey DR, Divertie MB, Didier EP. Preoperative pulmonary preparation of patients with chronic obstructive pulmonary disease: a prospective study. Chest. 1979 Aug;76(2):123-9. doi: 10.1378/chest.76.2.123. PMID 456049
- [Background] Svensson LG, Hess KR, Coselli JS, Safi HJ, Crawford ES. A prospective study of respiratory failure after high-risk surgery on the thoracoabdominal aorta. J Vasc Surg. 1991 Sep;14(3):271-82. PMID 1880835
- [Background] Arozullah AM, Daley J, Henderson WG, Khuri SF. Multifactorial risk index for predicting postoperative respiratory failure in men after major noncardiac surgery. The National Veterans Administration Surgical Quality Improvement Program. Ann Surg. 2000 Aug;232(2):242-53. doi: 10.1097/00000658-200008000-00015. PMID 10903604
- [Background] Hilmi IA, Damian D, Al-Khafaji A, Planinsic R, Boucek C, Sakai T, Chang CC, Kellum JA. Acute kidney injury following orthotopic liver transplantation: incidence, risk factors, and effects on patient and graft outcomes. Br J Anaesth. 2015 Jun;114(6):919-26. doi: 10.1093/bja/aeu556. Epub 2015 Feb 10. PMID 25673576
- [Background] Salvalaggio PR, Felga GE, Afonso RC, Ferraz-Neto BH. Early allograft dysfunction and liver transplant outcomes: a single center retrospective study. Transplant Proc. 2012 Oct;44(8):2449-51. doi: 10.1016/j.transproceed.2012.08.002. PMID 23026617
- [Background] Olthoff KM, Kulik L, Samstein B, Kaminski M, Abecassis M, Emond J, Shaked A, Christie JD. Validation of a current definition of early allograft dysfunction in liver transplant recipients and analysis of risk factors. Liver Transpl. 2010 Aug;16(8):943-9. doi: 10.1002/lt.22091. PMID 20677285
- [Background] Tapuria N, Kumar Y, Habib MM, Abu Amara M, Seifalian AM, Davidson BR. Remote ischemic preconditioning: a novel protective method from ischemia reperfusion injury--a review. J Surg Res. 2008 Dec;150(2):304-30. doi: 10.1016/j.jss.2007.12.747. Epub 2008 Jan 22. PMID 19040966
- [Background] Przyklenk K, Whittaker P. Genesis of remote conditioning: action at a distance--'hypotheses non fingo'? J Cardiovasc Med (Hagerstown). 2013 Mar;14(3):180-6. doi: 10.2459/JCM.0b013e328358c8eb. PMID 22964648
- [Background] McCafferty K, Forbes S, Thiemermann C, Yaqoob MM. The challenge of translating ischemic conditioning from animal models to humans: the role of comorbidities. Dis Model Mech. 2014 Dec;7(12):1321-33. doi: 10.1242/dmm.016741. PMID 25481012
- [Background] Ali ZA, Callaghan CJ, Lim E, Ali AA, Nouraei SA, Akthar AM, Boyle JR, Varty K, Kharbanda RK, Dutka DP, Gaunt ME. Remote ischemic preconditioning reduces myocardial and renal injury after elective abdominal aortic aneurysm repair: a randomized controlled trial. Circulation. 2007 Sep 11;116(11 Suppl):I98-105. doi: 10.1161/circulationaha.106.679167. PMID 17846333
- [Background] Zarbock A, Schmidt C, Van Aken H, Wempe C, Martens S, Zahn PK, Wolf B, Goebel U, Schwer CI, Rosenberger P, Haeberle H, Gorlich D, Kellum JA, Meersch M; RenalRIPC Investigators. Effect of remote ischemic preconditioning on kidney injury among high-risk patients undergoing cardiac surgery: a randomized clinical trial. JAMA. 2015 Jun 2;313(21):2133-41. doi: 10.1001/jama.2015.4189. PMID 26024502
- [Background] Kottenberg E, Thielmann M, Bergmann L, Heine T, Jakob H, Heusch G, Peters J. Protection by remote ischemic preconditioning during coronary artery bypass graft surgery with isoflurane but not propofol - a clinical trial. Acta Anaesthesiol Scand. 2012 Jan;56(1):30-8. doi: 10.1111/j.1399-6576.2011.02585.x. Epub 2011 Nov 21. PMID 22103808
- [Background] MacAllister R, Clayton T, Knight R, Robertson S, Nicholas J, Motwani M, Veighey K. REmote preconditioning for Protection Against Ischaemia-Reperfusion in renal transplantation (REPAIR): a multicentre, multinational, double-blind, factorial designed randomised controlled trial. Southampton (UK): NIHR Journals Library; 2015 May. Available from http://www.ncbi.nlm.nih.gov/books/NBK294375/ PMID 26020087
- [Background] Gonzalez NR, Hamilton R, Bilgin-Freiert A, Dusick J, Vespa P, Hu X, Asgari S. Cerebral hemodynamic and metabolic effects of remote ischemic preconditioning in patients with subarachnoid hemorrhage. Acta Neurochir Suppl. 2013;115:193-8. doi: 10.1007/978-3-7091-1192-5_36. PMID 22890668
- [Background] Li S, Ma C, Shao G, Esmail F, Hua Y, Jia L, Qin J, Ren C, Luo Y, Ding Y, Borlongan CV, Ji X. Safety and Feasibility of Remote Limb Ischemic Preconditioning in Patients With Unilateral Middle Cerebral Artery Stenosis and Healthy Volunteers. Cell Transplant. 2015;24(9):1901-11. doi: 10.3727/096368914X683520. Epub 2014 Jul 30. PMID 25198862
- [Background] Koch S, Katsnelson M, Dong C, Perez-Pinzon M. Remote ischemic limb preconditioning after subarachnoid hemorrhage: a phase Ib study of safety and feasibility. Stroke. 2011 May;42(5):1387-91. doi: 10.1161/STROKEAHA.110.605840. Epub 2011 Mar 17. PMID 21415404
- [Background] Rehni AK, Shri R, Singh M. Remote ischaemic preconditioning and prevention of cerebral injury. Indian J Exp Biol. 2007 Mar;45(3):247-52. PMID 17373368
- [Background] Section 2: AKI Definition. Kidney Int Suppl (2011). 2012 Mar;2(1):19-36. doi: 10.1038/kisup.2011.32. No abstract available. PMID 25018918
- [Background] Feng S, Goodrich NP, Bragg-Gresham JL, Dykstra DM, Punch JD, DebRoy MA, Greenstein SM, Merion RM. Characteristics associated with liver graft failure: the concept of a donor risk index. Am J Transplant. 2006 Apr;6(4):783-90. doi: 10.1111/j.1600-6143.2006.01242.x. PMID 16539636
- [Background] Meng R, Asmaro K, Meng L, Liu Y, Ma C, Xi C, Li G, Ren C, Luo Y, Ling F, Jia J, Hua Y, Wang X, Ding Y, Lo EH, Ji X. Upper limb ischemic preconditioning prevents recurrent stroke in intracranial arterial stenosis. Neurology. 2012 Oct 30;79(18):1853-61. doi: 10.1212/WNL.0b013e318271f76a. Epub 2012 Oct 3. PMID 23035060
- [Background] Bilgin-Freiert A, Dusick JR, Stein NR, Etchepare M, Vespa P, Gonzalez NR. Muscle microdialysis to confirm sublethal ischemia in the induction of remote ischemic preconditioning. Transl Stroke Res. 2012 Jun;3(2):266-72. doi: 10.1007/s12975-012-0153-1. Epub 2012 Apr 10. PMID 24323782
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of participants, 94, reflects the enrolled subjects, 31 + historical controls, 63.
Groups:
- Historical Control Cohort: Matched historical controls
Period: Overall Study
Arm/Group | Remote Ischemic Conditioning (RIC) Group | Historical Control Cohort
Started | 51 | 70
Screening | 51 | 70
Enrollment | 31 | 63
Protocol Completion | 22 | 63
Follow up | 31 | 63
Analyses (One in RIC cohort excluded in analyses of graft related outcomes since no transplant was performed) | 30 | 63
Completed | 31 | 63
Not Completed | 20 | 7
Not completed — Failed screening | 20 | 7

BASELINE CHARACTERISTICS:
Groups:
- Remote Ischemic Conditioning (RIC) Cohort: Subjects received remote ischemic conditioning
- Historical Control Cohort: Historical control subjects received liver transplants in an earlier period
- Total: Total of all reporting groups
Arm/Group | Remote Ischemic Conditioning (RIC) Cohort | Historical Control Cohort | Total
Number analyzed (Participants) | 31 | 63 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 56 | 82
  >=65 years | 5 | 7 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55.0 [51.0 to 63.0] | 56.0 [49.0 to 61.0] | 56 [48 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 26 | 32
  Male | 25 | 37 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 11 | 34 | 45
  More than one race | 6 | 6 | 12
  Unknown or Not Reported | 9 | 14 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 63 | 94

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Completing Entire Intervention Protocol
Description: Proportion of enrolled liver recipients that complete all 6 remote ischemic conditioning (RIC) interventions.
Time Frame: Pre-op - Post-op day 4
Population: Participants enrolled to receive RIC during transplant and the initial four post-transplant days and who receive all 6 RIC interventions.Subjects in historical control cohort chosen as described above
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remote Ischemic Conditioning (RIC) Group
Number analyzed (Participants) | 31
percentage of participants | 70.96 [54.04 to 87.89]

2. Secondary Outcome: Intervention-related Pain Score
Description: Median intervention-related pain score during each of the post-operative interventions, in extubated patients who are able to communicate. Using the Numerical Rating Scale (NRS, Ferrieira-Valente MA PAIN Volume 152, 2011), patients were asked to rate their pain following the intervention on a scale of 0-10 with 0 being no pain experienced to 10 as the maximum pain felt.
Time Frame: Post-op days 1-4
Population: Unintubated subjects were asked to rate intervention-related pain on a scale from 0-10 for each of the postoperative interventions. The maximum pain score obtained from each subject was recorded and the median score for all subjects was calculated. Scale range from 0 - 10 with 10 indicating highest sensation of pain.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Remote Ischemic Conditioning (RIC) Group
Number analyzed (Participants) | 23
scores on a scale | 5 [0 to 9]

3. Secondary Outcome: Withdrawal of Consent Due to Pain
Description: - Withdrawal of consent due to discomfort/pain in the lower extremity
Time Frame: Pre-op - Post-op day 7
Population: Participants who withdrew consent due to pain from RIC intervention.
Measure: Number; unit: participants
Groups:
- Historical Control Cohort: Subjects in this cohort were chosen via retrospective record review, and selected applying the same inclusion and exclusion criteria as in the RIC cohort. They were chosen consecutively in revere-chronological order that began at the start of the study date. Target ratio of RIC:Controls was 1:2. No matching was performed for age, sex, and model for end stage liver disease (MELD) score.
Arm/Group | Remote Ischemic Conditioning (RIC) Group | Historical Control Cohort
Number analyzed (Participants) | 31 | 63
participants | 6 | 0

4. Secondary Outcome: Percentage of Participants Who Developed Early Allograft Dysfunction (EAD)
Description: Percentage of participants who developed Early Allograft Dysfunction (EAD) which is defined as:
  * Aspartate Transaminase (AST) or Alanine Transaminase (ALT)> 2,000 U/L at any point within the first seven post-transplant days, or
  * Total Bilirubin (TB) > 10 mg/dL on postoperative day 7,or
  * International Normalized Ratio (INR)> 1.6 on postoperative day 7.
Time Frame: Post-op days 0-7
Population: Denominator for this and other postoperative outcomes except death and complications was 30 due to the exclusion of subject who died prior to transplantation
Measure: Number; unit: percentage of participants
Groups:
- Historical Control Cohort: Historical matched recipient controls
Arm/Group | Remote Ischemic Conditioning (RIC) Group | Historical Control Cohort
Number analyzed (Participants) | 30 | 63
percentage of participants | 23.3 | 39.68

5. Secondary Outcome: Percentage of Participants Who Developed Prolonged Respiratory Insufficiency (PRI)
Description: Percentage of Participants who developed Prolonged Respiratory Insufficiency (PRI) defined as:
  * Ventilator support for >2 postoperative days after transplant, or
  * Reintubation after extubation, within 7 days of transplant. Patients who require brief re-intubation for an endoscopic, radiologic, or surgical procedure would not be considered to have PRI if they are extubated within 2 days of the end of the procedure.
Time Frame: Post-op days 0-7
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Remote Ischemic Conditioning (RIC) Group | Historical Control Cohort
Number analyzed (Participants) | 30 | 63
percentage of participants | 33.3 | 28.57

6. Secondary Outcome: Percentage of Participants Who Developed Acute Kidney Injury (AKI) Stages 2 or 3
Description: Percentage of participants who developed Acute Kidney Injury (AKI)
  Based on Kidney Disease - Improving Global Outcomes (KDIGO) criteria, AKI criteria are:
  Stage 2:
  - 2.0-2.9 fold rise in serum creatinine from baseline
  Stage 3:
  * > 3.0 fold rise in serum creatinine from baseline, or
  * Serum creatinine of > 4.0 mg/dL, with an acute (<48 hours) increase of 0.3 mg/dL in serum creatinine or subacute (< 7 days) increase in serum creatinine of 0.5 mg/dL, or
  * Initiation of renal replacement therapy.
Time Frame: Post-op days 0-7
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Remote Ischemic Conditioning (RIC) Group | Historical Control Cohort
Number analyzed (Participants) | 30 | 63
percentage of participants | 20.0 | 25.86

7. Secondary Outcome: Time to Dialysis Discontinuation
Description: In patients who are receiving dialysis pre-op, time to discontinuation of dialysis, if occurring within 90 days of transplantation.
Time Frame: Post-op days 0-90
Population: Time to discontinuation of dialysis
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Remote Ischemic Conditioning (RIC) Group | Historical Control Cohort
Number analyzed (Participants) | 1 | 4
days | 2 [2 to 2] | 15.5 [10.25 to 19]

8. Secondary Outcome: Presence of Clavien-Dindo Grade IIIb or Higher Complications
Description: Percentage of patients with Clavien-Dindo >/= grade III b complications (Dindo D, Demartines N, Clavien P, Annals of Surgery 2004).
  The Clavien-Dindo Complications grade ranges from Grade I (Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgetics, diuretics and electrolytes and physiotherapy. This grade also includes wound infections opened at the bedside) to Grade V (Death). Grade IIIb would be any intervention requiring general anesthesia.
Time Frame: Post-op days 0-30
Measure: Number; unit: percentage of participants
Arm/Group | Remote Ischemic Conditioning (RIC) Group | Historical Control Cohort
Number analyzed (Participants) | 30 | 63
percentage of participants | 51.1 | 47.62

9. Secondary Outcome: Clavien-Dindo Grade IIIb or Higher - Number of Complications
Description: In patients with Clavien-Dindo >/= IIIb complications, number of such complications per patient.
Time Frame: Post-op days 0-30
Measure: Median (Inter-Quartile Range); unit: Complications
Arm/Group | Remote Ischemic Conditioning (RIC) Group | Historical Control Cohort
Number analyzed (Participants) | 31 | 63
Complications | 1 [0 to 3] | 0 [0 to 2]

10. Secondary Outcome: Intensive Care Unit (ICU) Length of Stay (LOS)
Description: Number of days in ICU post-transplant. Starting at post-op day 0 and ending on the calendar date that the patient is transferred out of ICU, dies, or post-op day 90, whichever is soonest.
Time Frame: Post-op days 0 up to 90 days
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Remote Ischemic Conditioning (RIC) Group | Historical Control Cohort
Number analyzed (Participants) | 30 | 63
days | 3.5 [2 to 8] | 4 [3 to 6]

11. Secondary Outcome: Hospital LOS
Description: Number of days in hospital post-transplant. Starting at post-op day 0 and ending on the calendar date that the patient is leaves the hospital, dies, or post-op day 90, whichever is soonest.
Time Frame: Post-op days 0 up to 90 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Remote Ischemic Conditioning (RIC) Group | Historical Control Cohort
Number analyzed (Participants) | 30 | 63
days | 13 [8 to 33] | 10 [7 to 15]

12. Secondary Outcome: Liver Allograft Survival
Description: Percentage of patients with functioning allograft at 90 days post-transplant
Time Frame: Post-op day 90
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Remote Ischemic Conditioning (RIC) Group | Historical Control Cohort
Number analyzed (Participants) | 30 | 63
percentage of participants | 90 | 98.41

13. Secondary Outcome: Patient Survival
Description: Percentage of patients alive at 90 days post-transplant
Time Frame: Post-op day 90
Measure: Number; unit: percentage of participants
Arm/Group | Remote Ischemic Conditioning (RIC) Group | Historical Control Cohort
Number analyzed (Participants) | 31 | 63
percentage of participants | 90.32 | 98.41

14. Secondary Outcome: Number of Subjects Not Completing Intervention Protocol
Description: Number of subjects that received fewer than 6 interventions,.
Time Frame: Pre-op - Post-op day 4
Population: Number of subjects who completed < 6 interventions
Measure: Number; unit: participants
Arm/Group | Remote Ischemic Conditioning (RIC) Group
Number analyzed (Participants) | 31
participants | 9

ADVERSE EVENTS:
Time Frame: Adverse events will be tracked for the first 30 days post-transplant.
Description: In addition to the clinical.trials. gov definitions, adverse events will be monitored related to the RIC intervention:
  Withdrawal of consent due to discomfort/pain in the lower extremity. Any other adverse event considered by the primary clinical team to be related to the RIC intervention.
Arm/Group | Remote Ischemic Conditioning (RIC) Group | Historical Control Cohort
All-Cause Mortality (participants affected / at risk) | 3/31 | 1/63
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/63
Other Adverse Events (participants affected / at risk) | 6/31 | 0/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remote Ischemic Conditioning (RIC) Group (N=31) | Historical Control Cohort (N=63)
Primary Non-Function of liver (Hepatobiliary disorders) | 1 (1) | 0 (0) — One subject experienced primary non-function between interventions 3 and 4 and did not receive further interventions
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remote Ischemic Conditioning (RIC) Group (N=31) | Historical Control Cohort (N=63)
Pain due to intervention (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) — Pain due to application of the RIC intervention was reported by the participants on a pain scale from 0-10 with 10 being the highest sensation of pain.

LIMITATIONS AND CAVEATS:
Two modifications resulted in a smaller number of subjects. Number of cycles, the duration of each cycle and the number of postoperative interventions were not addressed. Lack of randomization led to historical cohort to evaluate some outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT02635347/Prot_000.pdf
  • Informed Consent Form (2015-09-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT02635347/ICF_001.pdf
  • Statistical Analysis Plan (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT02635347/SAP_002.pdf